CLINICAL TRIAL: NCT04994080
Title: A Multi-center, Randomized, Double-blind, Parallel Grouping, Placebo-controlled Phase 3 Study to Assess the Efficacy and Safety of Paricalcitol Soft Capsules in the Treatment of Secondary Hyperparathyroidism in Subjects With Stage 3 and Stage 4 Chronic Kidney Disease
Brief Title: A Study to Assess the Efficacy and Safety of Paricalcitol in the Treatment of Chronic Kidney Disease With Secondary Hyperparathyroidism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-PLGHC-301
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-07

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Intervention Model Description: A multi-center, randomized, double-blind, parallel grouping, placebo-controlled phase 3 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A/B (Experimental)
  Interventions: Drug: Paricalcitol
- Treatment group C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol QD Treatment
  Arms: Treatment group A/B
Drug: Placebo — Placebo QD or TIW
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of Paricalcitol for secondary hyperparathyroidism with stage 3 and stage 4 chronic kidney disease in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Under care of physician at least 2 months for CKD
2. Not on active Vitamin D and Calcimimetic therapy for at least 4 weeks prior
3. If taking phosphate binders, on a stable regimen at least 4 weeks prior
4. For entry into Pretreatment Phase:

   iPTH at least 120 pg/mL GFR of 15-60 mL/min and no dialysis expected for at least 6 months
5. For entry into Treatment Phase:

Average of 2 consecutive iPTH values of at least 150 pg/mL, taken at least 1 day apart (all values not less than 120 pg/mL) 2 consecutive corrected serum calcium levels between 8.0-10.0 mg/dL 2 consecutive serum phosphorus levels of not more than 5.2 mg/mL

Exclusion Criteria:

1. Subjects who had Primary hyperparathyroidism;
2. Subjects with a history of acute renal failure;
3. Subjects with chronic gastrointestinal disease or severe liver disease with clinical symptoms;
4. Subjects with a history of unstable angina, grade III or IV congestive heart failure, and/or clinically meaningful arrhythmia;
5. Subjects with serum albumin < 30g/L, serum hemaoglobin < 85g/L, or serum transaminase higher than 2.5 times the upper limit of nomal;
6. Subjects with a history of malignancy;
7. Subjects who plan to undergo surgery during the study period;
8. Subjects with a history active granulomatous diseases;
9. Subject with a history of alcohol abuse and drug abuse;
10. Human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab) or Treponema pallidum antibody (TP-Ab) are positive;
11. Subjects who are allergic to the test drug and its ingredients or excipients;
12. Subjects who combined with systemic or systemic diseases that are not suitable for clinical trials;
13. Subjects who have participated in clinical trials of other drugs or devices;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with >30% decrease from basline at least twice in mean iPTH during the efficacy assessment phase. | 0-24 weeks

SECONDARY OUTCOMES:
The value of iPTH for each visit | 0-24 weeks
The change from baseline of iPTH for each visit | 0-24 weeks
The change percentage of iPTH for each visit; | 0-24 weeks
The proportion of subjects whose iPTH has been reduced by more than 30% from baseline at least 4 consecutive times; | 0-24 weeks
The change value in blood calcium from baseline; | 0-24 weeks
The change value in blood phosphorus from baseline; | 0-24 weeks
The change value in calcium-phosphorus product from baseline; | 0-24 weeks
The change value of 24-hour urine calcium from baseline; | 0-24 weeks
The change value of 24-hour urine phosphorus from baseline; | 0-24 weeks
The change value of 24-hour creatinine clearance rate from baseline; | 0-24 weeks
The change value of eGFR from baseline; | 0-24 weeks
The change value in urine calcium/creatinine ratio from baseline. | 0-24 weeks